CLINICAL TRIAL: NCT01507961
Title: Comparison of Soft and Hard Tissue Thickness in the Anterior Regions of the Upper and Lower Jaws Taken From CBCT Versus Clinical Measurements
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0229-11-HMO
Record Dates: First submitted 2012-01-08; First posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2011-12

CONDITIONS: Soft and Hard Tissue Biotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: there is a positive correlation between tissue thickness measured from CBCT and clinical measurements.

ELIGIBILITY:
Inclusion Criteria:

* 100 subject who have done a CT

Exclusion Criteria:

* periodontal surgery in anterior regions, medications which effect the gingiva

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 subjects who have done a CT
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-02